CLINICAL TRIAL: NCT04912180
Title: Apple Respiratory Study: A Prospective Study of Apple Watch-based Detection of Respiratory Viral Illness in Greater Seattle, WA
Brief Title: Apple Respiratory Study
Acronym: ARS
Status: Terminated | Type: Observational
Why Stopped: Study endpoints no longer feasible.
Sponsor: Apple Inc. (Industry)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00050502; STUDY00011439/ ARS-2020-001 (Other: University of Washington Human Subjects Division)
Record Dates: First submitted 2021-05-04; First posted 2021-06-03 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Acute Respiratory Infection; Coronavirus Infection; Influenza
MeSH Terms: conditions — Coronavirus Infections; Influenza, Human

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Apple Respiratory Study, a collaboration between researchers at Apple Inc. (the "Study Sponsor" or "Sponsor") and the Seattle Flu Study team at the University of Washington (UW) (the "UW Study Team"), is a prospective, longitudinal cohort, low risk Study to collect certain data from Apple Watch and iPhone to determine whether such data can detect physiologic and non-physiologic changes in individuals associated with respiratory illnesses due to influenza, SARS-CoV-2 and other respiratory pathogens (the "Study").

DETAILED DESCRIPTION:
Initial Screening and Study enrollment will begin in 2021 among adults residing in the Greater Seattle area. Participants will be recruited and driven to the online Study Website managed by UW. If determined to be eligible following completion of the Prescreen Consent and an initial eligibility assessment via REDCap, potential participants will be asked to review and, if interested in participation, to complete the Main Study Consent via REDCap, as well as to engage in enrollment procedures across both REDCap and the Apple Research app. Redcap will be used for prescreening, enrollment survey, and kit activation survey. Participants will use the Apple Research app to complete onboarding surveys, weekly symptom surveys, illness follow-up surveys, and monthly lifestyle surveys. These surveys will help the investigators learn about onset of respiratory symptoms as well as sick contacts, flu and/or COVID-19 vaccination and risk factors for illness. Participants will also receive an Apple Watch to capture certain sensor data-which, along with iPhone sensor data, will be correlated with symptom onset and symptom trajectory. If a participant experiences an acute respiratory illness (ARI), defined as at least one respiratory symptom for at least 24 hours, that individual will be asked to complete a symptom onset survey and self-collect an anterior nasal swab, which will be sent to UW Laboratory Medicine for analysis. Participants will be able to access their COVID swab test results using a secure web portal. Additionally, individuals who test positive or inconclusive for SARS-CoV-2 will be notified via phone by the UW Study Team and given instructions as defined by and in accordance with state, local, and national public health guidance.

ELIGIBILITY:
Inclusion Criteria:

To participate in this Study, individuals must:

* Have access to an iPhone 6s or later with compatible iOS as defined by the Apple App Store.
* Have regular and reliable internet access
* Be willing to comply with all Study procedures, including regular use of the Apple Watch (daytime and nighttime), complete the REDCap and Apple Research app surveys, share data from required Apple Watch and iPhone sensors, and perform self-collected nasal swabs
* Be able to read and comprehend English
* Be able to provide informed consent without the use of a legally authorized representative
* Have a permanent mailing address in the greater Seattle area where Study materials can be mailed
* Be at least 22 years old at the time of consent

Exclusion Criteria:

To participate in this Study, individuals must not:

* Have previously tested positive for SARS-CoV-2 via PCR or antibody test
* Currently be enrolled in University of Washington Husky Coronavirus Testing, Household Observation Study, or any other Seattle Flu Study sub-Study
* Have received any vaccine for COVID-19 or have an upcoming appointment for at least one dose of any COVID-19 vaccine prior to Study consent

Individuals also may be excluded from the Study once target participant counts have been achieved for certain demographics, comorbidity groups, and/or residence based on zip code

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Study aims to enroll up to 1000 adults. We estimate that we will detect approximately 70 laboratory confirmed influenza cases and 40 laboratory confirmed SARS-CoV-2 cases based on estimated event rate incidences.
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Symptomatic individuals that self-report ARI and have a laboratory-confirmed positive test for SARS-CoV-2 and/or influenza within 72 hours | Up to 6 months
  Proportion of symptomatic individuals that self-report ARI and have a laboratory-confirmed positive test for SARS-CoV-2 and/or influenza by self-swab within 72 hours of symptom onset.

SECONDARY OUTCOMES:
Self-report ARI and positive test for SARS-CoV-2 and/or influenza within 7 days | Up to 6 months
  Proportion of symptomatic individuals that self-report ARI and have a laboratory-confirmed positive test for SARS-CoV-2 and/or influenza by self-swab within 7 days of symptom onset.
Self-report ARI and test positive for other ARI within 7 days of symptom onset | Up to 6 months
  Proportion of symptomatic individuals that self-report ARI and test positive for another respiratory pathogen by self-swab within 7 days of symptom onset
Onset of ARI event | Up to 6 months
  Onset of ARI event defined as date and time of first self-reported symptoms (Day 0)
Hand washing Sessions | Up to 6 months
  Completed hand washing sessions per week as detected by Apple Watch
Measure of Heart Rate | Up to 6 months
  Measure of Heart Rate in Heart Beats per minute
Measure of Heart Rate Variability | Up to 6 months
  Measure of Heart Rate Variability in the standard deviation in the time interval between heart beats in milliseconds over variable periods of time.
Measure of Blood Oxygen | Up to 6 months
  Measure of Blood oxygen or oxygen saturation -percentage of hemoglobin in your red blood cells carrying oxygen (taken from Apple Watch)
Nasal swab sample that returns with no pathogens (viral and bacterial) on the panel | Up to 6 months
  Pathogen-negative ARI (pathogen not detected by laboratory testing; "pathogen negative ARI" could be due to chronic respiratory diseases, viral clearance, or inadequate sample collection)
RNaseP and viral CRT values | Up to 6 months
  RNaseP and viral CRT values for laboratory-confirmed virus positive ARI episodes
Duration of viral shedding and viral loads | Up to 6 months
  Duration of viral shedding and viral loads in COVID-positive patients as assessed by four swabs collected over two weeks of follow-up
ECG Reports | Up to 6 months
  Wrist-based Electrocardiogram (ECG) from smart watch containing time-series representation of the measured voltage corresponding to heart function over 30 second measurement periods.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Chu, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
The individual study data will not be shared beyond the investigative team, and only available to the sponsor in coded form. These details are outlined in the study protocol.